CLINICAL TRIAL: NCT01453101
Title: A Phase II Study of Allogeneic Hematopoietic Stem Cell Transplantation for Multiple Myeloma Using a Conditioning Regimen of Fludarabine, Melphalan, and Bortezomib
Brief Title: Allogeneic Hematopoietic Stem Cell Transplantation for Multiple Myeloma
Acronym: Flu-Mel-Vel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO1261
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine phosphate; Melphalan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludarabine, Melphalan, Bortezomib (Other)
  Interventions: Drug: Fludarabine monophosphate, melphalan, Bortezomib

INTERVENTIONS:
Drug: Fludarabine monophosphate, melphalan, Bortezomib — * Fludarabine will be administered at a dose of 30/mg/m2 IV daily for 4 days starting on transplant day -5.
  * Melphalan will be administered at a dose of 140 mg/m2 on transplant day-2
  * Bortezomib will be administered by rapid IV push at a dose of 1.6mg/m2 on days-4 and -1. The bortezomib should be given at least 20 hours after the melphalan.
  Other Names: Fludara; Phenylalanine Mustard; Velcade

SUMMARY:
The hypothesis for this study is that the regimen consisting of fludarabine, melphalan and bortezomib improves the progression free survival and the response rate compared to historical controls of fludarabine and melphalan alone.

DETAILED DESCRIPTION:
Multiple myeloma is the second most prevalent blood cancer (10%) after non-hodgkin's lymphoma. It represents approximately 1% of all cancers and 2% of all cancer deaths. Although the peak age of onset of multiple myeloma is 70 years of age, recent statistics indicate both increasing incidence and earlier age of onset.

The historical control 2-year progression-free survival (PFS) is assumed to be 35%. The proposed therapy of fludarabine, melphalan and bortezomib is expected to improve the PFS by 20%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma
* Have a suitable related or unrelated donor
* Age ≥18 but <70 yrs
* KPS of ≥70%
* Recovery from complications of previous therapies

Exclusion Criteria:

* Diagnosis other than multiple myeloma
* Chemotherapy or radiotherapy within 21 days of initiating treatment in this study
* Prior dose-intense therapy requiring HSC support within 56 days of initiating treatment in this study
* Uncontrolled bacterial, viral, fungal or parasitic infections
* Uncontrolled CNS metastases
* Known amyloid deposition in heart
* Organ dysfunction
* LVEF <40% or cardiac failure not responsive to therapy
* FVC, FEV1, or DLCO <50% of predicted and/or receiving supplementary continuous oxygen
* Evidence of hepatic synthetic dysfunction, or total bilirubin >2x or AST >3x ULN
* Measured creatinine clearance <20 ml/min
* Sensory peripheral neuropathy grade 4 within 14 days of enrollment
* Karnofsky score <70% unless a result of bone disease directly caused by myeloma
* Life expectancy limited by another co-morbid illness
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Female subject is pregnant or breast-feeding (women) or unwilling to use acceptable birth control methods (men or women) for twelve months after treatment. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Documented hypersensitivity to fludarabine or melphalan or to bortezomib, boron or mannitol or any components of the formulation
* Patients unable or unwilling to provide consent
* Patient has a sustained platelet count of <30 x 10 9/L within 14 days before enrollment
* Patient has a sustained absolute neutrophil count of <1.0 x10 9/L within 14 days before enrollment
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fludarabine, Melphalan, Bortezomib: Fludarabine monophosphate, melphalan, Bortezomib: •Fludarabine will be administered at a dose of 30/mg/m2 IV daily for 4 days starting on transplant day -5.
  * Melphalan will be administered at a dose of 140 mg/m2 on transplant day-2
  * Bortezomib will be administered by rapid IV push at a dose of 1.6mg/m2 on days-4 and -1. The bortezomib should be given at least 20 hours after the melphalan.
Period: Overall Study
Arm/Group | Fludarabine, Melphalan, Bortezomib
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine, Melphalan, Bortezomib
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 56 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The main primary endpoint of this study is two-year progression free survival. Patients are considered a failure with respect to PFS if they die or experience disease progression or relapse. The time to this event is the time from transplantation to relapse/progression, initiation of non-protocol anti-myeloma therapy, or death from any cause. Subjects alive without confirmed disease progression will be censored at the time of last disease evaluation. Deaths without progression are treated as failures no matter when they occur.
Time Frame: Subjects will be followed for progression-free survival for at least 36 months
Measure: Median (Full Range); unit: Months
Arm/Group | Fludarabine, Melphalan, Bortezomib
Number analyzed (Participants) | 54
Months | 16.7 [0.3 to 61.1]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS): Defined as time from the first dose of administration to death from any cause
Time Frame: Up to 3 years
Measure: Number; unit: percentage
Arm/Group | Fludarabine, Melphalan, Bortezomib
Number analyzed (Participants) | 54
percentage | 42

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate: Defined as the composite endpoint of response to treatment which includes Complete Response (CR), Partial Response (PR), stable disease (SD) as defined in International Response Criteria.
  International Myeloma Working Group Response Criteria for Multiple Myeloma:
  CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow PR: > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h SD: Not meeting criteria for CR, VGPR, PR, or progressive disease
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Fludarabine, Melphalan, Bortezomib
Number analyzed (Participants) | 54
Participants | 45

ADVERSE EVENTS:
Time Frame: Collected for 3 years post transplant per patient
Arm/Group | Fludarabine, Melphalan, Bortezomib
All-Cause Mortality (participants affected / at risk) | 27/54
Serious Adverse Events (participants affected / at risk) | 29/54
Other Adverse Events (participants affected / at risk) | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fludarabine, Melphalan, Bortezomib (N=54)
Rectal Hemmorhage (Gastrointestinal disorders) | 1
hemorrhoidal rectal bleed (Gastrointestinal disorders) | 1
fever (General disorders) | 10
infection/sepsis/URI (Infections and infestations) | 29
Renal Failure (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Graft versus Host Disease (Immune system disorders) | 9
Diarrhea (Gastrointestinal disorders) | 3
Intractable Migraine (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Respiratory Distress/Fluid Overload (Respiratory, thoracic and mediastinal disorders) | 1
Decreased Visual Acuity (Eye disorders) | 1
Multisystem Failure (General disorders) | 3
Nausea and Vomiting (Gastrointestinal disorders) | 1
Metapneumovirus Infection (Respiratory, thoracic and mediastinal disorders) | 3
Veno Occlusive Disease (Vascular disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Hemolytic Anemia (Vascular disorders) | 1
Epidural Tumor (Nervous system disorders) | 1
Progressive Disease (General disorders) | 7
GI Disorder (Gastrointestinal disorders) | 2
Confusion (General disorders) | 2
Hyponatremia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
GI Pain (Gastrointestinal disorders) | 1
Diabetic Ketoacidosis (Endocrine disorders) | 1
Cerebral Edema (Nervous system disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 1
Malnutrition (Gastrointestinal disorders) | 1
Fall (General disorders) | 1
Abdominal Wall Cellulitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT01453101/Prot_SAP_000.pdf